CLINICAL TRIAL: NCT05478213
Title: Ventricular Tachycardia Substrate Mechanisms Revealed by Local Repolarization and Conduction Parameters
Brief Title: Ventricular Tachycardia Mechanisms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Neal Bhatia, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003571; 2024P008207 (Other: Emory IRB)
Record Dates: First submitted 2022-06-28; First posted 2022-07-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular tachycardia ablation
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Monophasic Action Potential (MAP) Catheter (Experimental): Participants undergoing ventricular tachycardia ablation per standard of care will also have cellular action potential of the ventricular myocardium assessed with the MAP catheter.
  Interventions: Device: Monophasic Action Potential (MAP) Catheter

INTERVENTIONS:
Device: Monophasic Action Potential (MAP) Catheter — The EasyMap catheter is a temporary quadripolar catheter for recording monophasic action potentials and for intracardiac pacing. During a standard of care VT ablation, the MAP catheter will be used to study cellular action potential of the ventricular myocardium, which cannot be done on traditional catheters. The catheter is placed on the myocardium (similar to other traditional catheters) and a recording signal is transmitted to the workstation. Using the MAP catheter the will not interrupt or distort any of the standard treatment procedures.
  Other Names: EasyMap catheter

SUMMARY:
The purpose of this study is to understand why certain hearts have ventricular arrhythmias and help identify areas of the heart that cause arrhythmias. There is still a significant gap in understanding why ventricular arrhythmias occur. This study will examine the electrical properties of the heart tissue to understand how these arrhythmias occur, and hopefully identify areas that might lead to ventricular arrhythmias. The hope is that studying this might be able to improve outcomes during ventricular tachycardia (VT) ablations.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) ablation remains the cornerstone treatment for drug refractory VT. Previous studies have reported success rate of VT ablation ranging from 23 to 49%. Despite improvements in mapping and catheter technology, there is a high recurrence rate and numerous patients who fail VT ablation.

Reasons for failure in VT ablation include the inability to identify critical areas of myocardium responsible for VT and hemodynamic instability of VT during mapping. Several studies have attempted to study electrical properties of cardiac tissues to identify potential circuits in sinus rhythm avoid mapping during unstable VT. This includes mapping fractionated electrical potentials, isochronal late activation mapping (ILAM), and ablation of low voltage regions. However, these techniques have yielded modest improvement in success rates with poor specificity of identifying important regions.

Monophasic action potentials (MAP) demonstrate cellular action potential of the myocardium. Recent evidence suggests that changes in MAP morphology can predict sudden cardiac death by ventricular arrhythmias. However, cellular activation has not been studied in VT. The researchers of this study propose that MAP signals can better elucidate electrophysiological characteristics of the myocardium, and thus identify sites critical to VT.

During a standard of care VT ablation, the researchers will use the MAP catheter to study cellular action potential of the ventricular myocardium, which cannot be done on traditional catheters. The design of this catheter is similar to other diagnostic catheters that are currently used for VT ablation. The MAP catheter is a bipolar catheter, two with electrical poles at the distal tip. The catheter is placed on the myocardium (similar to other traditional catheters) and a recording signal is transmitted to the workstation. Using the MAP catheter the will not interrupt or distort any of the standard treatment procedures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic cardiomyopathy
* Single or dual chamber implantable cardioverter-defibrillator (ICD)

Exclusion Criteria:

* Non-Ischemic cardiomyopathy
* Contraindication to catheter ablation
* Severe peripheral arterial disease or medical condition that prohibit arterial access
* Ventricular tachycardia (VT) or sudden cardiac arrest (SCA) within 30 days of acute coronary syndrome or within 90 days of coronary revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Waveform Morphology | During ablation on Day 1
  Identification of sites that are critical to reentry of ventricular tachycardia from bystander sites will be performed by analyzing local ventricular activation. Local ventricular action is assessed with waveform morphology and is measured in voltage (mV). The normal range is >3 mV bipolar and >8.3 mV unipolar.
Conduction Velocity | During ablation on Day 1
  Identification of sites that are critical to reentry of ventricular tachycardia from bystander sites will be performed by analyzing electrophysiological properties. Electrophysiological properties are assessed with conduction velocity, measured in meters per second (m/s).

SECONDARY OUTCOMES:
Identify mechanisms of slowed conduction at ILAM | During ablation on Day 1
  The mechanisms responsible for slowed conduction at sites that are critical to ventricular tachycardia using monophasic action potential signals will be examined.
Identify surrogate markers | During ablation on Day 1
  Surrogate markers for monophasic action potential tracings will be compared to conventional mapping catheters.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Bhatia, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No